CLINICAL TRIAL: NCT03681769
Title: Developing Brain Stimulation as a Treatment for Chronic Pain in Opiate Dependent
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00078668; UG3DA048506 (Other Grant/Funding Number: National Institute on Drug Abuse); R21DA044503 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-24 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain; Opiate Dependence; Lower Back Pain
Keywords: Transcranial Magnetic Stimulation; Dorsolateral Prefrontal Cortex; Medial Prefrontal Cortex; Brain Stimulation
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, sham-controlled study will parametrically evaluate the longitudinal effects of 16 days of rTMS to the DLPFC (Aim 1) or the MPFC (Aim 2) on self-reported pain and the brain's response to pain. This will be done in a cohort of patients recruited from Medical University of South Carolina clinics and the outer community with chronic lower back pain that have been using prescription opiates for 3 or more months without adequate pain relief. Participants will be randomized to receive TMS to the DLPFC, MPFC, or sham (50% at each site), using a Latin square randomization. Resting state connectivity will be collected along with data from a standardized thermal pain paradigm wherein individuals are exposed to pain and instructed to try to "control' the pain. Quantitative Pain Testing will be collected 12 times. MRI data will be collected 3 times: before the 1st visit of TMS, before the 12th visit of TMS, and before the 16th visit of TMS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data for this randomized, double-blind, sham-controlled study (behavioral assessments, functional MRI measurements) will be acquired by the members of the Dr. Hanlon's lab, including graduate students and research specialists. These individuals will also perform data under the guidance of the PI. Manuscript composition will be led by the PI, with the assistance of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Intermittent Theta Burst Stimulation (iTBS) to the left dlPFC (Experimental): For intermittent theta burst stimulation (iTBS) (Aim 1), participants will receive 20 trains of stimulation over the dlPFC (middle frontal gyrus) (F3) (each train: 3 pulse bursts presented at 5 hertz, 15 pulses/sec for 2 sec, 8 sec rest, 200 pulses/train; 110% resting motor threshold, MagPro; 600 pulses total) using a figure 8 coil (Coil Cool-B65 A/P).
  Interventions: Device: iTBS to the left dlPFC
- Sham iTBS to the left dlPFC (Sham Comparator): The MagVenture MagPro system has an integrated, active sham which passes current through two surface electrodes placed on the scalp. The electrodes will be placed on the left frontalis muscle for all sessions. A patient identification card will randomize participants to receive either real or sham stimulation. This system maintains blinding by a gyroscope in the coil which indicates to the clinical staff whether the coil should be rotated up or down for this participant once the card is entered into the machine. One side of the coil is active, the other is sham. The integrity of the double-blind procedure will be assessed by asking the patients and study personnel rate their confidence regarding whether they thought they received real or sham (scale 1-10).
  Interventions: Device: Sham iTBS to the left dlPFC
- cTBS to the mPFC (Experimental): For continuous theta burst stimulation (Aim 2), participants will receive 1 train of stimulation over the left frontal pole (FP1) (each train: 3 pulse bursts presented at 5 hertz, 15 pulses/sec for 40 sec, 600 pulses/train, 110% resting motor threshold, MagPro; 600 pulses total) using a figure 8 coil (Coil Cool-B65 A/P). This protocol has been shown to attenuate the mPFC and striatum in cocaine dependent individuals in the past (61-63) and has been more effective than 1200 or 1800 pulses of cTBS in attenuating depression (The time between the end of the TBS procedures and the beginning of the behavioral assessments, as well as the scalp-to-cortex distance (which effects the actual TMS dose given to the cortex) will be compiled and used as covariates in subsequent analyses.
  Interventions: Device: cTBS to the mPFC
- Sham cTBS to the mPFC (Sham Comparator): The MagVenture MagPro system has an integrated, active sham which passes current through two surface electrodes placed on the scalp. The electrodes will be placed on the left frontalis muscle for all sessions. A patient identification card will randomize participants to receive either real or sham stimulation. This system maintains blinding by a gyroscope in the coil which indicates to the clinical staff whether the coil should be rotated up or down for this participant once the card is entered into the machine. One side of the coil is active, the other is sham. The integrity of the double-blind procedure will be assessed by asking the patients and study personnel rate their confidence regarding whether they thought they received real or sham (scale 1-10).
  Interventions: Device: Sham cTBS to the mPFC

INTERVENTIONS:
Device: iTBS to the left dlPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the Universal Serial Bus (USB) key).
  Arms: Intermittent Theta Burst Stimulation (iTBS) to the left dlPFC
Device: Sham iTBS to the left dlPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham iTBS to the left dlPFC
Device: cTBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key)
  Arms: cTBS to the mPFC
Device: Sham cTBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham cTBS to the mPFC

SUMMARY:
Effective control of chronic pain is a top priority in the United States, as approximately 10% of adults have severe chronic pain - most of which is chronic lower back pain (CLBP). However, despite the advances in neuroscience over the past 20 years, chronic pain is still largely treated with opiate narcotics, much as was done in the Civil War. In addition to the high abuse liability and dependence potential, only 30-40% of chronic pain patients declare they receive satisfactory (>50%) relief from their pain through pharmacological treatment. In these patients a common clinical practice is to escalate the dose of opiates as tolerance develops - which unfortunately has contributed to escalation in opiate overdose deaths, a resurgence of intravenous heroin use, and $55 billion in societal costs. Consequently there is a critical need for new, treatments that can treat pain and reduce reliance on opiates in individuals with chronic pain.

Aim 1. Evaluate repetitive Transcranial Magnetic Stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC) as a tool to dampen pain and the engagement of the Pain Network. Hypothesis 1: DLPFC TMS will attenuate the baseline brain response to pain (Pain Network activity) and increase activity in the Executive Control Network (ECN) when the patient is given instructions to 'control' the pain.

Aim 2. Evaluate Medial Prefrontal Cortex (MPFC) rTMS as a tool to dampen pain and the engagement of the Pain Network. Hypothesis 1: MPFC TMS will also attenuate the baseline brain response to pain (Pain Network activity) but will not effect the ECN or the Salience Network (SN) when the patient is given instructions to 'control' the pain.

DETAILED DESCRIPTION:
The goal of this proposal is to evaluate two novel non-invasive brain stimulation strategies to mitigate pain and the brain's response to pain in CLBP patients. Transcranial Magnetic Stimulation (TMS), can induce long term potentiation (LTP-like) and long term depression (LTD-like) effects on brain activity in a frequency dependent manner. The investigators have previously demonstrated that LTP-like TMS to the dorsolateral prefrontal cortex (DLPFC, a node in the Executive Control Network (ECN)) can decrease perceived pain and corresponding Blood Oxygen Level Dependent (BOLD) signal in the "Pain Network'. The Pain Network is an expansion of the Salience Network (SN; insula, dorsal anterior cingulate) which includes the thalamus and somatosensory cortex. The analgesic effects of DLPFC TMS can be blocked by naloxone - suggesting that the analgesic effects of LTP-like DLPFC TMS are opiate mediated. Additionally, DLPFC TMS delivered postoperatively leads to less patient administered morphine use (PCA-pump) in the hospital and less opiate use in the outpatient setting. These data all suggest that LTP-like DLPFC TMS is a promising candidate for treating pain.

An alternative strategy is to apply LTD-like stimulation to the medial prefrontal cortex (LTD-like mPFC rTMS. This strategy is based on the understanding of functional neural architecture, wherein the SN is modulated by two other core networks: the ECN and the default mode network (DMN). As stated above, it is possible to attenuate activity in the SN through LTP-like TMS to the DLPFC, a node in the ECN. It is also possible to attenuate the SN through LTD-like TMS to the ventral medial prefrontal cortex (a node in the DMN). The proposed study will be the first to employ a randomized, double-blind, sham-controlled design to parametrically evaluate the longitudinal effects of 16 days of rTMS to the DLPFC (Aim 1) or the MPFC (Aim 2) on self-reported pain and the brain's response to pain. This will be done in a cohort of patients recruited from the community as well as Medical University of South Carolina clinics with chronic lower back pain that may or may not be using prescription opiates for 3 or more months without adequate pain relief. Participants will be randomized to receive rTMS to the DLPFC (10Hz), MPFC (cTBS), or sham (50% at each site), using a Latin square randomization. Resting state connectivity will be collected along with data from a standardized thermal pain paradigm wherein individuals are exposed to pain and instructed to try to "control' the pain. MRI data will be collected 3 times: before the 1st day of TMS, after the 12th day of TMS, and before the 16th day of TMS (the last day administered).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 (to maximize participation)
* Currently using prescription opiates
* Able to read and understand questionnaires and informed consent.
* Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold)
* Does not have metal objects in the head/neck.
* Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.
* Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

* Any psychoactive illicit substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine Carboxy-Tetrahydrocannabinol levels.
* Meets Diagnostic and Statistical Manual of Mental Disorders IV criteria for current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder or organic mental disorder.
* Has current suicidal ideation or homicidal ideation.
* Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for Attention Deficit Hyperactivity Disorder.
* Females of childbearing potential who are pregnant (by urine human chorionic gonadotropin level), nursing, or who are not using a reliable form of birth control.
* Has current charges pending for a violent crime (not including driving under the influence related offenses).
* Does not have a stable living situation.
* Suffers from chronic migraines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex: For intermittent theta burst stimulation (iTBS) (Aim 1), participants will receive 20 trains of stimulation over the motor cortex (each train: 3 pulse bursts presented at 5 hertz, 15 pulses/sec for 2 sec, 8 sec rest, 200 pulses/train; 110% resting motor threshold, MagPro; 600 pulses total) using a figure 8 coil (Coil Cool-B65 A/P).
  iTBS to the Motor Cortex: This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the Universal Serial Bus (USB) key).
Period: Overall Study
Arm/Group | Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC | Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex: For intermittent theta burst stimulation (iTBS) (Aim 1), participants will receive 20 trains of stimulation over the dlPFC (middle frontal gyrus) (F3) (each train: 3 pulse bursts presented at 5 hertz, 15 pulses/sec for 2 sec, 8 sec rest, 200 pulses/train; 110% resting motor threshold, MagPro; 600 pulses total) using a figure 8 coil (Coil Cool-B65 A/P).
  iTBS to the Motor Cortex: This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the Universal Serial Bus (USB) key).
- Total: Total of all reporting groups
Arm/Group | Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC | Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (14.2) | 57.7 (10.9) | 53.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Quantitative Pain Testing Following Active TMS Compared to Baseline
Description: Based on pilot data, the investigators expect an interaction between treatment (DLPFC or MC rTMS) and time (Before vs. After rTMS) on reported painfulness using a quantitative sensory testing technique that determines thermal pain threshold.
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: Change from Baseline (degrees C)
Arm/Group | Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC | Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex
Number analyzed (Participants) | 11 | 11
Change from Baseline (degrees C) | 1.4 (.3) | .3 (.15)
Statistical Analysis 1: Comparison: Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC vs Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex; Test type: Equivalence — Non-equivalence determined by p<.05; p = .83, Mixed Models Analysis — No site X time interaction (F12,270 = 0.614, p = 0.830)

2. Secondary Outcome: Change in Patient Reported Pain and Discomfort
Description: The investigators expect reductions in self reported pain assessment via a numeric pain rating scale when comparing active vs sham. Pain rating values will be assessed and reported through the duration of the study. Numeric Rating Scale (NRS) for pain has a range of 0 to 10 where 0=no pain/discomfort and 10=worst pain/discomfort imaginable. Higher scores mean more pain/discomfort.
Time Frame: Patient reported pain/discomfort at 16 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC | Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex
Number analyzed (Participants) | 11 | 11
score on a scale | 5.3 (2.4) | 5.9 (2.0)
Statistical Analysis 1: Comparison: Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC vs Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex; Test type: Other; p = .53, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to 16 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Intermittent Theta Burst Stimulation (iTBS) to the Left dlPFC | Intermittent Theta Burst Stimulation (iTBS) to the Motor Cortex
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03681769/Prot_SAP_000.pdf